CLINICAL TRIAL: NCT02185040
Title: A Pilot, Phase 2, Randomized, Placebo-Controlled, Double-Blind, Study To Evaluate Efficacy, Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Pharmacogenetics of CC-220 In Subjects With Systemic Lupus Erythematosus
Brief Title: A Pilot Study of CC-220 to Treat Systemic Lupus Erythematosus.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-220-SLE-001
Record Dates: First submitted 2014-07-07; First posted 2014-07-09 (Estimated); Results first posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus, Systemic Lupus, SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — iberdomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- CC-220 0.3mg Every Other Day (QOD) (Experimental): Part 1: CC-220 0.3mg capsules by mouth every other day (QOD)
  Interventions: Drug: CC-220
- CC-220 0.3mg Every Day (QD) (Experimental): * Part 1: CC-220 0.3mg capsules by mouth every day (QD)
  * ATEP: CC-220 0.3 mg capsules by mouth every day (QD)
  Interventions: Drug: CC-220
- CC-220 0.6mg/0.3mg alternating dose QD (Experimental): * Part 1: CC-220 0.6 mg and 0.3mg capsules PO on alternating days
  * ATEP:CC-220 0.6 mg and 0.3 mg capsules PO on alternating days
  Interventions: Drug: CC-220
- CC-220 0.6mg QD (Experimental): Part 1: CC-220 0.6mg capsules by mouth QD
  Interventions: Drug: CC-220
- Placebo QD (Placebo Comparator): Part 1: Identically matching placebo capsules PO QD
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CC-220 — 0.3 mg oral capsules once every other day with or without food
  Arms: CC-220 0.3mg Every Other Day (QOD)
Drug: CC-220 — Subjects will receive 0.3 mg oral capsules every day with or without food
  Arms: CC-220 0.3mg Every Day (QD)
Drug: CC-220 — CC-220 oral capsules 0.6 mg and 0.3 mg on alternating days with or without food
  Arms: CC-220 0.6mg/0.3mg alternating dose QD
Drug: CC-220 — CC-220 oral capsule 0.6 mg QD with or without food
  Arms: CC-220 0.6mg QD
Drug: Placebo — Matching oral placebo daily
  Arms: Placebo QD

SUMMARY:
The purpose of this study is to determine whether CC-220 is effective for the treatment of skin, joint and serological manifestations of systemic lupus erythematosus.

DETAILED DESCRIPTION:
The study consists of 2 parts. Part 1 is a randomized, double-blind, placebo controlled, ascending dose study to evaluate the safety and tolerability of CC-220 in SLE subjects.

Subject participation in Part 1 consists of 3 phases:

* Pre-treatment Screening Phase: up to 28 days prior to the first dose of the investigational product (IP)
* Treatment Phase: up to 84 days
* Observation Phase: 84 day post-treatment A total of approximately 40 subjects will be randomized into 4 dose groups with a 4:1 ratio of CC-220 (0.3 mg every other day [QOD], 0.3 mg everyday [QD], 0.6 mg and 0.3 mg on alternating days, and 0.6 mg QD) or matching placebo. In each dosing arm, 8 subjects will receive active drug and 2 subjects will receive placebo. The Treatment Phase will be up to 84 days in duration for all dose groups. Subjects who discontinue IP early and all subjects who complete the 84 day treatment phase will enter into the Observational Follow-up Phase for an 84 day period. A subject will be permitted to reduce their dose one time during Part 1 of the study.

Part 2 is the Active Treatment Extension Phase (ATEP) which is an extension to evaluate the long-term efficacy and safety/tolerability of CC-220 in SLE subjects who completed Part 1 of the study. Subjects who complete the Treatment Phase of Part 1 of the study will be eligible to receive CC-220 in the ATEP for up to 2 years. All subjects who participate in the ATEP will receive either 0.3 mg QD or 0.6 mg and 0.3 mg QD on alternating days. Subjects who terminate the Treatment Phase of Part 1 early will not be eligible for entry into the ATEP.

Subject participation consists of two phases:

* Active Treatment Extension Phase: Up to 2 years
* Observational Follow-up Phase: One month

ELIGIBILITY:
Inclusion Criteria:

Part 1

* The subject has an established diagnosis of systemic lupus erythematosus (SLE) as defined by the 1997 Update of the 1982 ACR Revised Criteria for Classification of SLE at screening. The diagnosis is fulfilled provided that at least 4 criteria are met.
* Disease history of SLE ≥ 6 months at baseline
* Females of childbearing potential (FCBP) must:

  * Have two negative pregnancy tests as verified by the study doctor prior to starting study therapy. She must agree to ongoing pregnancy testing during the course of the study, and after end of study therapy. This applies even if the subject practices true abstinence from heterosexual contact.
  * Either commit to true abstinence from heterosexual contact (which must be reviewed on a monthly basis) or agree to use, and be able to comply with, effective contraception without interruption, 28 days prior to starting IP, during the study therapy (including dose interruptions), and for 28 days after discontinuation of study therapy.
* Male subjects must:

  * Must practice true abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 28 days following IP discontinuation, even if he has undergone a successful vasectomy.
  * If the subject is using oral corticosteroids, the daily dose must be less than or equal to 10 mg of prednisone or equivalent during the study; the dose must be stable over the 4 weeks preceding screening and throughout the study.
  * All subjects taking hydroxychloroquine, chloroquine and/or quinacrine during the study must have documentation of a normal ophthalmologic examination performed within 1 year of the Baseline Visit.
  * For subjects not taking corticosteroids, or antimalarials, the last dose (in case of previous use) must be at least 4 weeks prior to screening.

ATEP

* Male or female 18 years of age or older
* Understand and voluntarily sign an ICD prior to the initiation of any study related assessments/procedures
* Able to adhere to the study visit schedule and other protocol requirements. Pregnancy
* Females of childbearing potential (FCBP) must:

  * Have two negative pregnancy tests as verified by the study doctor prior to starting study therapy. She must agree to ongoing pregnancy testing during the course of the study, and after end of study therapy. This applies even if the subject practices true abstinence* from heterosexual contact.
  * Either commit to true abstinence* from heterosexual contact (which must be reviewed on a monthly basis) or agree to use, and be able to comply with, effective contraception without interruption, 28 days prior to starting IP, during the study therapy (including dose interruptions), and for 28 days after discontinuation of study therapy.
* Male subjects must:

  - Practice true abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 28 days following IP discontinuation, even if he has undergone a successful vasectomy. True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
* Male subjects must agree not to donate semen or sperm during therapy and for at least 90 days following the discontinuation of IP.
* All subjects must:

  * Understand that the IP could have potential teratogenic risk
  * Agree to abstain from donating blood while taking IP and for 28 days following discontinuation of the IP
  * Agree not to share IP with another person
  * Other than the subject, FCBP and males able to father a child should not handle the IP or touch the capsules unless gloves are worn
  * Be counseled about pregnancy precautions and risks of fetal exposure as described in the Pregnancy Prevention Plan. Concomitant Medications
* If the subject is using oral corticosteroids, the daily dose must be less than or equal to 10 mg of prednisone or equivalent during the study; the dose must be stable over the 4 weeks preceding randomization and throughout the study.
* All subjects taking hydroxychloroquine, chloroquine or quinacrine during the study must have documentation of a normal ophthalmologic examination performed within 1 year of the Baseline Visit.
* For subjects not taking corticosteroids the last dose (in case of previous use) must be at least 4 weeks prior to screening.

Exclusion Criteria

* The subject has been treated with intra-articular, intramuscular or IV pulse corticosteroids within 4 weeks of screening.
* The subject has received high dose oral prednisone (> 100 mg/day) within 4 weeks of screening.
* The subject has received cyclophosphamide, azathioprine or mycophenolate mofetil within 12 weeks of screening.
* The subject has participated in a clinical trial and has received an investigational product within 30 days, 5 pharmacokinetic half-lives or twice the duration of the biological effect of the investigational product (whichever is longer) prior to screening; OR participation in two or more investigational drug trials within 12 months of screening.
* Unstable lupus nephritis defined as: proteinuria > 1.0 g/24 hour /1.73 m2 OR eGFR of less than 60 mL/1.73 m2 CNS disease, including active severe CNS lupus (including seizures, psychosis, organic brain syndrome, cerebrovascular accident (CVA), cerebritis or CNS vasculitis) requiring therapeutic intervention within 6 months of screening.
* The subject has New York Heart Association (NYHA) Class III or IV congestive heart failure.
* Presence of hepatitis B surface antigen (HBsAG). Subjects may have a positive anti-hepatitis B core antibody (anti-HBc) if the anti-hepatitis B surface antibody (anti-HBs) is positive as well.
* Antibodies to hepatitis C at Screening.
* The subject has a known positive history of antibodies to human immunodeficiency virus (HIV) or HIV disease or acquired immune deficiency syndrome (AIDs).
* Has a history of an organ transplant (e.g., heart, lung, kidney, liver) or hematopoietic stem cell/marrow transplant.
* Malignancy or history of malignancy, except for:

  * treated (ie, cured) basal cell or squamous cell in situ skin carcinomas;
  * treated (ie, cured) cervical intraepithelial neoplasia (CIN) or carcinoma in situ of the cervix with no evidence of recurrence within 5 years of Screening
* Systemic bacterial infections requiring treatment with oral or injectable antibiotics, or significant viral or fungal infections, within 4 weeks of Screening. Any treatment for such infections must have been completed and the infection cured, at least 2 weeks prior to Screening and no new or recurrent infections prior to the Baseline visit.
* History of venous thrombosis or any thromboembolic events within 2 years of screening.
* Clinical evidence of significant unstable or uncontrolled acute or chronic disease not due to SLE (ie, cardiovascular, pulmonary, hematologic, gastrointestinal, hepatic, renal, neurological, malignancy, psychiatric or infectious disease) which in the opinion of the investigator could put the subject at undue risk or confound study results.
* Presence of active uveitis or any other clinically significant ophthalmological finding.
* History or current diagnosis of peripheral or radicular neuropathy. Any clinically significant abnormalities on ECG, which, in the opinion of the investigator would interfere with safe participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-09-16 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2018-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shimon Korish, M.D., Study Director — Celgene
Locations (35):
- United States (35):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Arthritis and Rheumatology Research, PLLC, Paradise Valley, Arizona
  - University of Arizona Clinical and Translational Science Research Center, Tucson, Arizona
  - UCSD Center for Innovative Therapy, La Jolla, California
  - Dermatology Research Associates, Los Angeles, California
  - East Bay Rheumatology Medical Group Inc., San Leandro, California
  - Clinical Science Institute, Santa Monica, California
  - Los Angeles Biomedical Research Institute at Harbor - UCLA, Torrance, California
  - Inland Rheumatology Clinical Trials, Upland, California
  - Vipul Joshi, MD, PA, dba Bay Area Arthritis and Osteoporosis, Brandon, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Advanced Medical Research, Atlanta, Georgia
  - Arthritis Research and Treatment Center, Stockbridge, Georgia
  - Northwestern Medical Group; Department of Dermatology, Chicago, Illinois
  - Northshore University Health System, Skokie, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Northwell Health / Division of Rheumatology, Lake Success, New York
  - Feinstein Institute For Medical Research, Manhasset, New York
  - NYU Langone Medical Center, New York, New York
  - Columbia Presbyterian Medical Center, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - DJL Clinical Research, Charlotte, North Carolina
  - MetroHealth Medical Systems, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - University of Pennsylvania Health Systems, Philadelphia, Pennsylvania
  - UMPC Lupus Center of Excellence, Pittsburgh, Pennsylvania
  - Low Country Rheumatology PA, Charleston, South Carolina
  - Austin Regional Clinic, Austin, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia
  - Seattle Arthritis Clinic, Seattle, Washington

REFERENCES:
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The multi-center study was conducted in the United States. Forty-two participants were enrolled at 11 study sites.
Pre-assignment Details: In part 1 of the study, participants were randomly assigned to 1 of 4 dose cohorts; within each cohort participants were randomized in a 4:1 ratio to receive iberdomide or placebo. Participants who completed the Part 1 treatment phase were eligible to receive iberdomide for up to 2 years in the active treatment extension phase (ATEP).
Groups:
- Part 1: Placebo: Participants received identically matching placebo capsules for up to 84 days during the Part 1 treatment phase.
- Part 1: Iberdomide 0.3 mg QOD: Participants received iberdomide 0.3 mg capsules every other day (QOD) for up to 84 days during Part 1 treatment phase.
- Part 1: Iberdomide 0.3 mg QD: Participants received 0.3 mg iberdomide capsules once a day (QD) for up to 84 days during the Part 1 treatment phase.
- Part 1: Iberdomide 0.6 mg/0.3 mg ALT Days: Participants received iberdomide 0.6 mg and 0.3 mg on alternating days (ALT QD) for up to 84 days during the Part 1 treatment phase.
- Part 1: Iberdomide 0.6 mg QD: Participants received 0.6 mg iberdomide capsules QD for up to 84 days during Part 1 treatment phase.
- ATEP: Iberdomide 0.3 mg QD: Participants originally assigned to the iberdomide 0.3 mg capsules QD or 0.3 mg Iberdomide capsules QOD or placebo cohorts (in these respective groups) in Part 1 treatment phase, were assigned 0.3 mg iberdomide capsules QD when entered into the active treatment extension phase (ATEP) and continued iberdomide 0.3 mg QD up to 2 years.
- ATEP: Iberdomide 0.6 mg/0.3 mg ALT Days: Participants originally assigned to the iberdomide 0.6 mg capsules QD or 0.6 mg iberdomide capsules alternating with 0.3 mg iberdomide capsules or placebo QD cohorts, (in these perspective groups) in Part 1 treatment phase, were assigned 0.3 mg iberdomide capsules on alternating days with 0.6 mg capsules when entered into the active treatment extension phase and continued for up to 2 years. Participants who were initially assigned to 0.6 mg iberdomide QD in Part 1 treatment phase, were assigned to 0.6 mg iberdomide QD up to protocol amendment 5 when the dose was reduced. Participants who received 0.6 mg iberdomide QD were assigned and analyzed with the 0.3/0.6 iberdomide ALT QD group in the ATEP.
Period: Part 1 Treatment Phase
Arm/Group | Part 1: Placebo | Part 1: Iberdomide 0.3 mg QOD | Part 1: Iberdomide 0.3 mg QD | Part 1: Iberdomide 0.6 mg/0.3 mg ALT Days | Part 1: Iberdomide 0.6 mg QD | ATEP: Iberdomide 0.3 mg QD | ATEP: Iberdomide 0.6 mg/0.3 mg ALT Days
Started | 8 | 8 | 8 | 9 | 9 | 0 | 0
Completed | 7 | 6 | 7 | 7 | 6 | 0 | 0
Not Completed | 1 | 2 | 1 | 2 | 3 | 0 | 0
Not completed — Miscellaneous | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 2 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Active Treatment Extension Phase
Arm/Group | Part 1: Placebo | Part 1: Iberdomide 0.3 mg QOD | Part 1: Iberdomide 0.3 mg QD | Part 1: Iberdomide 0.6 mg/0.3 mg ALT Days | Part 1: Iberdomide 0.6 mg QD | ATEP: Iberdomide 0.3 mg QD | ATEP: Iberdomide 0.6 mg/0.3 mg ALT Days
Started | 0 | 0 | 0 | 0 | 0 | 9 | 8
Completed | 0 | 0 | 0 | 0 | 0 | 6 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 3 | 7
Not completed — Miscellaneous | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) includes all participants who were randomized and received at least 1 dose of investigational product (IP). Participants were included in the treatment group to which they were randomized for the ITT analyses.
Groups:
- Part 1: Iberdomide 0.3 mg QD: Participants received 0.3 mg iberdomide capsules QD up to 84 days during the Part 1 treatment phase and remained on their assigned dose of 0.3 mg iberdomide capsules QD during ATEP up to 2 years.
- Part 1: Iberdomide 0.6 mg/0.3 mg ALT Days: Participants received iberdomide 0.6 mg capsules on alternating (ALT) days with 0.3 mg iberdomide capsules on alternating days up to 84 days during the Part 1 treatment phase and remained on their assigned dose of 0.3 mg iberdomide capsules ALT days with 0.6 mg capsules ALT days during the ATEP up to 2 years.
- Total: Total of all reporting groups
Arm/Group | Part 1: Placebo | Part 1: Iberdomide 0.3 mg QOD | Part 1: Iberdomide 0.3 mg QD | Part 1: Iberdomide 0.6 mg/0.3 mg ALT Days | Part 1: Iberdomide 0.6 mg QD | Total
Number analyzed (Participants) | 8 | 8 | 8 | 9 | 9 | 42
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.8 (6.58) | 46.0 (8.62) | 48.0 (10.85) | 49.8 (13.07) | 47.2 (13.56) | 47.2 (10.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 7 | 8 | 9 | 39
  Male | 1 | 0 | 1 | 1 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 1 | 1 | 1 | 7
  Not Hispanic or Latino | 5 | 7 | 7 | 8 | 8 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 2 | 2 | 4 | 1 | 4 | 13
  White | 5 | 6 | 4 | 7 | 5 | 27
  Other | 0 | 0 | 0 | 1 | 0 | 1
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 33.029 (5.8922) | 30.119 (5.7386) | 36.426 (9.9918) | 27.012 (4.9291) | 28.553 (8.3143) | 30.873 (7.6362)
Cutaneous Lupus Area and Severity Index Activity Score (CLASI) Activity Score [Mean (Standard Deviation); unit: units on a scale] — The CLASI Activity Score ranges from 0 to 70 and is generated as: erythema scale = 0 (absent) to 3 (dark red; purple/violaceous/crusted/hemorrhagic) and scale/hypertrophy = 0 (absent) to 2 (verrucous/hypertrophic). Erythema and hypertrophy scores are assessed in 13 anatomical locations. The presence of mucous membrane lesions is scored on a scale of 0 (absent) to 1 (lesion), and hair loss is captured (1 = yes; 0 = no); nonscarring alopecia is scored: 0 (absent) to 3 (focal or patchy in ≥ 1 quadrant). Individual component scores are summed. Higher scores = greater cutaneous disease activity.
  units on a scale | 4.3 (5.90) | 17.6 (12.89) | 6.3 (9.07) | 8.4 (8.63) | 12.4 (16.48) | 9.8 (11.76)
Hybrid SELENA Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) [Mean (Standard Deviation); unit: Units on a Scale] — The SELENA SLEDAI score measures SLE disease activity of 24 lupus descriptors. Each descriptor receives a positive score if it is present over the previous assessment; a score of '0' = inactive disease; a positive score (from 1 - 8 is based on the importance of each descriptor in the total scoring) indicates disease activity. The SELENA SLEDAI score is the sum of all 24 descriptors' scores assessment period. The SELENA SLEDAI score can range from '0' to a maximum theoretical score of 105 (maximum SLE disease activity). The higher the SELENA SLEDAI score the greater of SLE disease activity.
  Units on a Scale | 6.8 (1.83) | 8.4 (4.07) | 5.5 (2.07) | 6.7 (3.16) | 5.7 (1.87) | 6.6 (2.79)
Physician's Global Assessment (PGA) [Mean (Standard Deviation); unit: Units on a Scale] — The PGA uses a visual analogue scale with ranges from 0 and 3 to indicate worsening of disease. The scoring was as follows:
  0 = none
  1. = mild disease
  2. = moderate disease
  3. = severe disease. The PGA is a physician administered instrument used to gauge a participant's overall state of health.
  Units on a Scale | 0.95 (0.518) | 1.50 (0.648) | 1.50 (0.614) | 1.22 (0.353) | 1.40 (0.598) | 1.31 (0.565)
Baseline Swollen Joint Count [Mean (Standard Deviation); unit: Swollen Joints] — Joint swelling was noted as "present" or "absent," with no quantitation of severity. Forty-four joints were evaluated for the presence or absence of swelling. The same evaluator performed the joint assessments for a given participant at the study site at each study visit. Population: Participants with least one swollen joint count.
  Swollen Joints
    number analyzed (Participants) | 5 | 5 | 6 | 8 | 4 | 28
    (all) | 4.0 (2.12) | 5.2 (2.28) | 7.0 (5.22) | 6.3 (2.49) | 4.0 (1.15) | 5.5 (3.11)
Baseline Tender Joint Count [Mean (Standard Deviation); unit: Joints] — Joint tenderness was noted as "present" or "absent," with no quantitation of severity. Forty-four joints were evaluated for the presence or absence of swelling. The same evaluator performed the joint assessments for a given participant at the study site at each study visit. Population: Participants with at least one tender joint count.
  Joints
    number analyzed (Participants) | 6 | 6 | 7 | 8 | 6 | 33
    (all) | 10.0 (7.21) | 7.3 (4.97) | 14.3 (9.66) | 16.9 (9.09) | 13.3 (11.29) | 12.7 (8.90)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) in Part 1 Treatment Phase
Description: A TEAE was defined as any adverse event (AE) that began or worsened on or after the start of IP up to 28 days after the last dose of IP or IP discontinuation date, whichever was later. Each participant was counted once for each applicable category. An IP-related TEAE was defined as a TEAE that the investigator considered to be of suspected relationship to IP. The severity of each adverse event and serious AE (SAE) was assessed by the investigator and graded based on a scale from mild - mild symptoms to severe AEs (non-serious or serious). A serious adverse event (SAE) was any AE which: • Resulted in death • Was life-threatening • Required inpatient hospitalization or prolongation of existing hospitalization • Resulted in persistent or significant disability/incapacity • Was a congenital anomaly/birth defect • Constituted an important medical event.
Time Frame: From the start of the first dose of IP until 28 days after the last dose or study discontinuation in Part 1; median treatment duration = 12.0 weeks for the placebo, 0.3 mg QOD and 0.3 mg iberdomide QD arms, 11.9 weeks for the 0.6/0.3 ALT and 0.6 cohorts.
Population: The safety population included all participants who were randomized and received at least 1 dose of IP. For all participants, this was the treatment group to which they were randomized.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1: Iberdomide 0.3 mg QD: Participants received 0.3 mg iberdomide capsules once a day for up to 84 days during the Part 1 treatment phase.
Arm/Group | Part 1: Placebo | Part 1: Iberdomide 0.3 mg QOD | Part 1: Iberdomide 0.3 mg QD | Part 1: Iberdomide 0.6 mg/0.3 mg ALT Days | Part 1: Iberdomide 0.6 mg QD
Number analyzed (Participants) | 8 | 8 | 8 | 9 | 9
Participants
  Any TEAE | 5 | 7 | 7 | 8 | 8
  Any IP-related TEAE | 1 | 2 | 2 | 4 | 6
  Any Severe TEAE | 1 | 0 | 0 | 1 | 2
  Any Serious TEAE | 2 | 0 | 0 | 1 | 1
  Any Serious IP-related TEAE | 0 | 0 | 0 | 0 | 1
  Any TEAE Leading to IP Interruption | 0 | 0 | 1 | 1 | 5
  Any TEAE Leading to IP Withdrawal | 1 | 0 | 0 | 2 | 3
  Any TEAE Leading to Death | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) in the Active Treatment Extension Phase
Description: A TEAE was defined as any adverse event (AE) that began or worsened on or after the start of IP through 28 days after the last dose of IP or IP discontinuation date, whichever was later. Each participant was counted once for each applicable category. An IP-related TEAE was defined as a TEAE that the investigator considered to be of suspected relationship to IP. The severity of each adverse event and serious AE (SAE) was assessed by the investigator and graded based on a scale from mild - mild symptoms to severe AEs (non-serious or serious). A serious adverse event (SAE) was any AE which: • Resulted in death • Was life-threatening • Required inpatient hospitalization or prolongation of existing hospitalization • Resulted in persistent or significant disability/incapacity • Was a congenital anomaly/birth defect • Constituted an important medical event.
Time Frame: From the date of the first dose of IP in the ATEP until 28 days after the last dose in the ATEP or study discontinuation; median duration of IP was 95.86 weeks for the 0.3 mg iberdomide QD cohort and 60.64 weeks for the 0.6 mg/0.3 mg ALT QD cohorts.
Population: The active treatment extension population included all participants who were enrolled into the ATEP and received at least 1 dose of IP.
Measure: Count of Participants; unit: Participants
Arm/Group | ATEP: Iberdomide 0.3 mg QD | ATEP: Iberdomide 0.6 mg/0.3 mg ALT Days
Number analyzed (Participants) | 9 | 8
Participants
  Any TEAE | 9 | 7
  Any IP-related TEAE | 2 | 5
  Any Severe TEAE | 0 | 5
  Any Serious TEAE | 0 | 4
  Any Serious IP-related TEAE | 0 | 0
  Any TEAE Leading to IP Interruption | 2 | 5
  Any TEAE Leading to IP Withdrawal | 1 | 4
  Any TEAE Leading to Death | 0 | 0

3. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time 0 to the Last Measurable Concentration (AUCt) of Iberdomide
Description: The area under the plasma concentration time curve (AUCt) was defined as area under the concentration-time curve from time zero to the last quantifiable time point, calculated by the linear trapezoidal rule when concentrations are increasing and the logarithmic trapezoidal method when concentrations are decreasing. Single and multiple-dose PK were collected in Part 1 of the study for all dose groups. Iberdomide reaches steady state within 7 days. PK collection on Day 29 was sufficient to understand PK once steady state was reached. As no dose adjustments were made in ATEP, further PK collection was not needed.
Time Frame: Pharmacokinetic (PK) blood samples were collected on Day 1 and Day 29 pre-dose (Time = 0 hours) and at 1, 2, 3, 4, between 6 and 8 hours and 24 hours after administration of IP.
Population: The PK population included all participants in the safety population with at least one non-missing plasma concentration datum available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part 1: Iberdomide 0.3 mg QOD | Part 1: Iberdomide 0.3 mg QD | Part 1: Iberdomide 0.6 mg/0.3 mg ALT Days | Part 1: Iberdomide 0.6 mg QD
Number analyzed (Participants) | 3 | 3 | 5 | 4
ng*h/mL
  Day 1 | 10.82 (17.9) | 11.29 (42.6) | 34.15 (45.5) | 38.73 (76.5)
  Day 29: number analyzed (Participants) | 3 | 3 | 4 | 3
  Day 29 | 13.34 (14.1) | 15.55 (1.8) | 24.85 (110.5) | 52.65 (82.4)

4. Secondary Outcome: Maximum Observed Concentration (Cmax) Of Iberdomide
Description: Maximum observed plasma concentration, obtained directly from the observed concentration versus time data. Single and multiple-dose PK were collected in Part 1 of the study for all dose groups. Iberdomide reaches steady state within 7 days. PK collection on Day 29 was sufficient to understand PK once steady state was reached. As no dose adjustments were made in ATEP, further PK collection was not needed.
Time Frame: Pharmacokinetic blood samples were collected on Day 1 and Day 29 at pre-dose (Time = 0 hours) and at 1, 2, 3, 4, between 6 and 8 hours and 24 hours after administration of IP.
Population: as for outcome 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1: Iberdomide 0.3 mg QOD | Part 1: Iberdomide 0.3 mg QD | Part 1: Iberdomide 0.6 mg/0.3 mg ALT Days | Part 1: Iberdomide 0.6 mg QD
Number analyzed (Participants) | 3 | 3 | 5 | 4
ng/mL
  Day 1: number analyzed (Participants) | 3 | 1 | 5 | 4
  Day 1 | 0.90 (41.3) | 0.64 (42.4) | 2.92 (50.6) | 2.35 (63.1)
  Day 29: number analyzed (Participants) | 3 | 3 | 4 | 3
  Day 29 | 1.02 (4.3) | 1.09 (1.8) | 2.37 (42.7) | 3.51 (51.7)

5. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) of Iberdomide
Description: Time to Cmax, obtained directly from the observed concentration versus time data. Single and multiple-dose PK were collected in Part 1 of the study for all dose groups. Iberdomide reaches steady state within 7 days. PK collection on Day 29 was sufficient to understand PK once steady state was reached. As no dose adjustments were made in ATEP, further PK collection was not needed.
Time Frame: as for outcome 4
Population: as for outcome 3
Measure: Median (Full Range); unit: days
Arm/Group | Part 1: Iberdomide 0.3 mg QOD | Part 1: Iberdomide 0.3 mg QD | Part 1: Iberdomide 0.6 mg/0.3 mg ALT Days | Part 1: Iberdomide 0.6 mg QD
Number analyzed (Participants) | 3 | 3 | 5 | 4
days
  Day 1: number analyzed (Participants) | 3 | 1 | 5 | 4
  Day 1 | 4.00 [2.0 to 4.0] | 6.00 [3.0 to 25.8] | 1.92 [0.95 to 4.0] | 4.01 [2.0 to 27.3]
  Day 29: number analyzed (Participants) | 3 | 3 | 4 | 3
  Day 29 | 4.00 [2.05 to 4.08] | 2.00 [2.0 to 3.05] | 3.00 [1.0 to 4.0] | 2.02 [1.1 to 3.1]

6. Secondary Outcome: Terminal Phase Half-Life (T1/2) Of Iberdomide
Description: Terminal phase half-life in plasma, calculated as [(In 2)/λz]. T1/2 half was only calculated when a reliable estimate for λz could be obtained. Single and multiple-dose PK were collected in Part 1 of the study for all dose groups. Iberdomide reaches steady state within 7 days. PK collection on Day 29 was sufficient to understand PK once steady state was reached. As no dose adjustments were made in ATEP, further PK collection was not needed.
Time Frame: as for outcome 4
Population: The Pharmacokinetic population included all participants in the safety population with at least one non-missing plasma concentration datum available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | Part 1: Iberdomide 0.3 mg QOD | Part 1: Iberdomide 0.3 mg QD | Part 1: Iberdomide 0.6 mg/0.3 mg ALT Days | Part 1: Iberdomide 0.6 mg QD
Number analyzed (Participants) | 1 | 3 | 5 | 4
days
  Day 1: number analyzed (Participants) | 1 | 1 | 3 | 2
  Day 1 | 7.50 (NA) — NA = Due to small sample size, the GCV% could not be calculated. | 10.25 (NA) — NA = Due to small sample size, the GCV% could not be calculated. | 7.96 (22.8) | 9.55 (0.2)
  Day 29: number analyzed (Participants) | 1 | 3 | 2 | 2
  Day 29 | 8.46 (NA) — NA = Due to small sample size, the GCV% could not be calculated. | 11.85 (4.1) | 9.39 (11.1) | 11.32 (4.8)

7. Secondary Outcome: Percentage of Participants Who Achieved ≥4 Points Reduction From Baseline in Hybrid Safety of Estrogens in Systemic Lupus Erythematosus National Assessment SLE Disease Activity Index Score (SELENA SLEDAI) During the ATEP by Time Point
Description: The SELENA SLEDAI score measures SLE disease activity through assessment of 24 lupus descriptors/manifestations. Each descriptor (clinical or lab values) receives a positive score if it is present over the previous assessment period; a score of '0' indicates inactive disease while a positive score (from 1 to 8 based on the relative importance of each descriptor in the total scoring) indicates disease activity. The SELENA SLEDAI score is the sum of all 24 descriptors' scores for the assessment period. The SELENA SLEDAI score can range from '0' (no SLE disease activity) to a maximum theoretical score of 105 (maximum SLE disease activity). The higher the SELENA SLEDAI score the greater of SLE disease activity.
Time Frame: Baseline to Weeks 1, 4, 12, 24, 36, 48, 60, 72, 84, 96 and follow-up at Week 100 during the ATEP.
Population: The active treatment extension population included all participants who were enrolled into the ATEP and received at least 1 dose of IP. The number analyzed at each time point includes participants with a baseline value >= 4 and non-missing post-baseline value.
Measure: Number; unit: Percentage of Participants
Arm/Group | ATEP: Iberdomide 0.3 mg QD | ATEP: Iberdomide 0.6 mg/0.3 mg ALT Days
Number analyzed (Participants) | 9 | 8
Percentage of Participants
  Week 1: number analyzed (Participants) | 7 | 8
  Week 1 | 0.0 | 12.5
  Week 4: number analyzed (Participants) | 7 | 7
  Week 4 | 0.0 | 14.3
  Week 12: number analyzed (Participants) | 6 | 7
  Week 12 | 66.7 | 0.0
  Week 24: number analyzed (Participants) | 6 | 5
  Week 24 | 83.3 | 20.0
  Week 36: number analyzed (Participants) | 6 | 4
  Week 36 | 66.7 | 0.0
  Week 48: number analyzed (Participants) | 6 | 5
  Week 48 | 50.0 | 20.0
  Week 60: number analyzed (Participants) | 6 | 5
  Week 60 | 33.3 | 20.0
  Week 72: number analyzed (Participants) | 5 | 3
  Week 72 | 80.0 | 0.0
  Week 84: number analyzed (Participants) | 5 | 2
  Week 84 | 80.0 | 0.0
  Week 96: number analyzed (Participants) | 5 | 1
  Week 96 | 40.0 | 0.0
  Week 100 Follow-Up: number analyzed (Participants) | 5 | 4
  Week 100 Follow-Up | 40.0 | 0.0

8. Secondary Outcome: Change From Baseline in the Hybrid Systemic Lupus Erythematosus Disease Activity Index (SELENA SLEDAI) During the ATEP by Time Point
Description: as for outcome 7
Time Frame: Baseline to Weeks 1, 4, 12, 24, 36, 48, 60, 72, 84, 96 and follow-up at Week 100 during the ATEP.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ATEP: Iberdomide 0.3 mg QD | ATEP: Iberdomide 0.6 mg/0.3 mg ALT Days
Number analyzed (Participants) | 9 | 8
Units on a Scale
  Week 1 | 0.2 (1.56) | -1.0 (2.39)
  Week 4: number analyzed (Participants) | 9 | 7
  Week 4 | 0.2 (1.56) | -1.7 (2.93)
  Week 12: number analyzed (Participants) | 8 | 7
  Week 12 | -1.8 (2.92) | -0.9 (1.07)
  Week 24: number analyzed (Participants) | 8 | 5
  Week 24 | -2.8 (2.60) | -1.2 (2.59)
  Week 36: number analyzed (Participants) | 7 | 4
  Week 36 | -3.1 (1.95) | 0.3 (2.06)
  Week 48: number analyzed (Participants) | 7 | 5
  Week 48 | -2.9 (1.95) | -1.0 (2.65)
  Week 60: number analyzed (Participants) | 7 | 5
  Week 60 | -2.6 (1.90) | -1.8 (4.02)
  Week 72: number analyzed (Participants) | 6 | 3
  Week 72 | -3.0 (1.67) | -1.3 (1.15)
  Week 84: number analyzed (Participants) | 6 | 2
  Week 84 | -3.0 (1.67) | -1.0 (1.41)
  Week 96: number analyzed (Participants) | 6 | 1
  Week 96 | -2.0 (1.79) | 0.0 (NA) — NA = Could not be calculated due to the low number of participants with available data.
  Week 100 Follow-Up: number analyzed (Participants) | 7 | 4
  Week 100 Follow-Up | -1.7 (2.43) | 0.3 (1.71)

9. Secondary Outcome: Change From Baseline in Swollen Joint Count During the ATEP by Time Point
Description: Joint swelling was noted as present or absent. Forty-four joints were assessed for swelling, including the sternoclavicular, acromioclavicular, shoulder, elbow, wrist, metacarpophalangeal (MCP), proximal interphalangeal (PIP), knee, ankle, and metatarsophalangeal (MTP) joints were included in this joint count.
Time Frame: Baseline to Weeks 1, 4, 12, 24, 36, 48, 60, 72, 84, 96 and follow-up at Week 100 during the ATEP.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | ATEP: Iberdomide 0.3 mg QD | ATEP: Iberdomide 0.6 mg/0.3 mg ALT Days
Number analyzed (Participants) | 9 | 8
Joints
  Week 1 | -1.2 (3.11) | -0.4 (0.74)
  Week 4: number analyzed (Participants) | 9 | 7
  Week 4 | -1.8 (2.99) | -0.6 (2.64)
  Week 12: number analyzed (Participants) | 8 | 7
  Week 12 | -2.6 (4.81) | -0.3 (0.95)
  Week 24: number analyzed (Participants) | 8 | 5
  Week 24 | -2.1 (5.84) | 1.2 (1.30)
  Week 36: number analyzed (Participants) | 7 | 5
  Week 36 | -3.9 (4.67) | -0.2 (2.17)
  Week 48: number analyzed (Participants) | 7 | 5
  Week 48 | -3.6 (5.35) | 0.6 (1.34)
  Week 60: number analyzed (Participants) | 7 | 5
  Week 60 | -2.6 (5.74) | 0.4 (1.52)
  Week 72: number analyzed (Participants) | 6 | 3
  Week 72 | -4.0 (5.10) | 0.7 (1.15)
  Week 84: number analyzed (Participants) | 6 | 2
  Week 84 | -4.2 (5.49) | 0.0 (0.00)
  Week 96: number analyzed (Participants) | 6 | 1
  Week 96 | -3.7 (5.75) | 0.0 (NA) — NA = Could not be calculated due to the low number of participants with available data.
  Week 100 Follow-Up: number analyzed (Participants) | 7 | 5
  Week 100 Follow-Up | -3.6 (5.26) | -0.4 (0.55)

10. Secondary Outcome: Change From Baseline in Tender Joint Count During the ATEP by Time Point
Description: Joint tenderness was noted as present or absent. Forty-four joints were assessed for swelling, including the sternoclavicular, acromioclavicular, shoulder, elbow, wrist, metacarpophalangeal (MCP), proximal interphalangeal (PIP), knee, ankle, and metatarsophalangeal (MTP) joints were included in this joint count.
Time Frame: Baseline to Weeks 1, 4, 12, 24, 36, 48, 60, 72, 84, 96 and follow-up at Week 100 during the ATEP.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | ATEP: Iberdomide 0.3 mg QD | ATEP: Iberdomide 0.6 mg/0.3 mg ALT Days
Number analyzed (Participants) | 9 | 8
Joints
  Week 1 | -0.9 (2.37) | -2.5 (4.63)
  Week 4: number analyzed (Participants) | 9 | 7
  Week 4 | -0.9 (3.76) | -2.0 (3.27)
  Week 12: number analyzed (Participants) | 8 | 7
  Week 12 | 0.5 (6.02) | -3.7 (7.67)
  Week 24: number analyzed (Participants) | 8 | 5
  Week 24 | -3.9 (4.19) | -3.6 (10.97)
  Week 36: number analyzed (Participants) | 7 | 5
  Week 36 | -5.1 (5.30) | -3.8 (9.65)
  Week 48: number analyzed (Participants) | 7 | 5
  Week 48 | -5.9 (6.99) | -3.0 (8.97)
  Week 60: number analyzed (Participants) | 7 | 5
  Week 60 | -5.6 (9.78) | -4.4 (10.99)
  Week 72: number analyzed (Participants) | 6 | 3
  Week 72 | -6.2 (6.59) | -6.7 (12.42)
  Week 84: number analyzed (Participants) | 6 | 2
  Week 84 | -7.3 (10.78) | 0.0 (0.00)
  Week 96: number analyzed (Participants) | 6 | 1
  Week 96 | -7.0 (7.92) | 0.0 (NA) — NA = Could not be calculated due to the low number of participants with available data.
  Week 100 Follow-Up: number analyzed (Participants) | 7 | 5
  Week 100 Follow-Up | -4.1 (3.63) | -1.4 (3.44)

11. Secondary Outcome: Percent Change From Baseline in Cutaneous Lupus Area and Severity Index (CLASI) Activity Score During the ATEP by Time Point
Description: The CLASI Activity Score ranges from 0 to 70. To generate the activity score erythema is scored on a scale of 0 (absent) to 3 (dark red; purple/violaceous/crusted/hemorrhagic) and scale/hypertrophy are scored on a scale of 0 (absent) to 2 (verrucous/hypertrophic). Both the erythema and scale/hypertrophy scores are assessed in 13 different anatomical locations. In addition, the presence of mucous membrane lesions is scored on a scale of 0 (absent) to 1 (lesion or ulceration), the occurrence of recent hair loss is captured (1=yes; 0=no) and nonscarring alopecia is scored on a scale of 0 (absent) to 3 (focal or patchy in more than one quadrant). To calculate the CLASI activity score, all scores for erythema, scale/hypertrophy, mucous membrane lesions and alopecia are added together. Composite scores are calculated by summing the individual component scores. The higher the score, the greater the cutaneous disease activity.
Time Frame: Baseline to Weeks 1, 4, 12, 24, 36, 48, 60, 72, 84, 96 and follow-up at Week 100 during the ATEP.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | ATEP: Iberdomide 0.3 mg QD | ATEP: Iberdomide 0.6 mg/0.3 mg ALT Days
Number analyzed (Participants) | 9 | 8
Percent Change
  Week 1: number analyzed (Participants) | 7 | 7
  Week 1 | -21.40 (40.529) | -13.35 (28.556)
  Week 4: number analyzed (Participants) | 7 | 6
  Week 4 | -32.13 (45.400) | -18.32 (58.924)
  Week 12: number analyzed (Participants) | 6 | 6
  Week 12 | -18.42 (68.423) | -36.46 (33.648)
  Week 24: number analyzed (Participants) | 6 | 4
  Week 24 | 13.54 (147.030) | -44.69 (24.366)
  Week 36: number analyzed (Participants) | 5 | 4
  Week 36 | -0.56 (116.911) | -43.98 (31.724)
  Week 48: number analyzed (Participants) | 5 | 4
  Week 48 | -46.97 (44.154) | -46.00 (22.343)
  Week 60: number analyzed (Participants) | 5 | 4
  Week 60 | -65.64 (40.889) | -47.51 (28.871)
  Week 72: number analyzed (Participants) | 4 | 2
  Week 72 | -55.13 (41.583) | -40.35 (9.924)
  Week 84: number analyzed (Participants) | 4 | 2
  Week 84 | -65.71 (24.535) | -32.46 (1.241)
  Week 96: number analyzed (Participants) | 4 | 1
  Week 96 | -75.38 (23.492) | -26.32 (NA) — NA = Could not be calculated due to the low number of participants with available data.
  Follow-Up Week 100: number analyzed (Participants) | 5 | 5
  Follow-Up Week 100 | -53.04 (39.635) | -18.82 (37.296)

12. Secondary Outcome: Change From Baseline in the Physician's Global Assessment (PGA) Score During the ATEP by Time Point
Description: The physician's global assessment was administered by the treating physician and was used to gauge the participants overall state of health. The instrument uses a visual analogue scale with scores between 0 and 3 to indicate worsening of disease. The scoring is as follows:
  * 0 = none
  * 1 = mild disease
  * 2 = moderate disease
  * 3 = severe disease
Time Frame: Baseline to Weeks 1, 4, 12, 24, 36, 48, 60, 72, 84, 96 and follow-up at Week 100 during the ATEP.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ATEP: Iberdomide 0.3 mg QD | ATEP: Iberdomide 0.6 mg/0.3 mg ALT Days
Number analyzed (Participants) | 9 | 8
Units on a Scale
  Week 1 | -0.08 (0.139) | -0.10 (0.245)
  Week 4: number analyzed (Participants) | 9 | 7
  Week 4 | -0.26 (0.510) | -0.17 (0.407)
  Week 12: number analyzed (Participants) | 8 | 7
  Week 12 | -0.15 (0.407) | -0.31 (0.389)
  Week 24: number analyzed (Participants) | 8 | 5
  Week 24 | -0.28 (0.686) | -0.20 (0.394)
  Week 36: number analyzed (Participants) | 7 | 5
  Week 36 | -0.30 (0.141) | -0.36 (0.590)
  Week 48: number analyzed (Participants) | 7 | 5
  Week 48 | -0.53 (0.556) | -0.26 (0.594)
  Week 60: number analyzed (Participants) | 7 | 5
  Week 60 | -0.37 (0.550) | -0.24 (0.498)
  Week 72: number analyzed (Participants) | 6 | 3
  Week 72 | -0.48 (0.471) | -0.23 (0.666)
  Week 84: number analyzed (Participants) | 6 | 2
  Week 84 | -0.57 (0.468) | -0.30 (0.707)
  Week 96: number analyzed (Participants) | 6 | 1
  Week 96 | -0.52 (0.595) | -0.20 (NA) — NA = Could not be calculated due to the low number of participants with available data.
  Follow-Up Week 100: number analyzed (Participants) | 7 | 5
  Follow-Up Week 100 | -0.21 (0.769) | 0.10 (0.354)

13. Secondary Outcome: Change From Baseline in the British Isles Lupus Assessment Group (BILAG) 2004 Global Score During the ATEP by Time Point
Description: The BILAG-2004 index measures clinical disease activity in systemic lupus erythematosus (SLE). A single alphabetic score (A through E) is used to denote disease severity for each of the 9 domains (constitutional, mucocutaneous, neuropsychiatric, musculoskeletal, cardiorespiratory, gastrointestinal, ophthalmic, renal, and hematologic). BILAG A represents the most active disease or severe disease; BILAG B represents intermediate activity or moderate disease; BILAG C represents stable mild disease; BILAG D represents organ system previously affected but now inactive; and BILAG E represents organ system never involved. The global BILAG score is the sum of a converted numerical score (A=9, B=3, C=1, D=0, E=0) over 9 domains. The theoretical range spans from 0 (no activity) to 13 active or severe disease activity BILAG. A higher score means more severe disease activity while a lower score means lower disease activity (or no disease activity for score of zero).
Time Frame: Baseline to Weeks 1, 4, 12, 24, 36, 48, 60, 72, 84, 96 and follow-up at Week 100 during the ATEP.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ATEP: Iberdomide 0.3 mg QD | ATEP: Iberdomide 0.6 mg/0.3 mg ALT Days
Number analyzed (Participants) | 9 | 8
Units on a Scale
  Week 1: number analyzed (Participants) | 8 | 7
  Week 1 | -0.5 (5.76) | 3.3 (5.38)
  Week 4: number analyzed (Participants) | 6 | 6
  Week 4 | 2.0 (7.04) | 0.7 (9.03)
  Week 12: number analyzed (Participants) | 5 | 6
  Week 12 | -2.2 (6.98) | 2.0 (6.03)
  Week 24: number analyzed (Participants) | 7 | 4
  Week 24 | -6.3 (6.55) | 3.0 (5.60)
  Global Score Week 36: number analyzed (Participants) | 7 | 5
  Global Score Week 36 | -7.3 (5.74) | 1.6 (9.13)
  Week 48: number analyzed (Participants) | 7 | 5
  Week 48 | -6.1 (7.84) | 1.4 (5.68)
  Week 60: number analyzed (Participants) | 7 | 5
  Week 60 | -6.3 (6.37) | 0.4 (4.83)
  Week 72: number analyzed (Participants) | 6 | 3
  Week 72 | -7.5 (4.46) | 4.3 (8.50)
  Week 84: number analyzed (Participants) | 6 | 2
  Week 84 | -7.8 (8.04) | -1.0 (1.41)
  Week 96: number analyzed (Participants) | 6 | 1
  Week 96 | -0.52 (0.595) | -0.20 (NA) — NA = Could not be calculated due to the low number of participants with available data.
  Follow-Up Week 100: number analyzed (Participants) | 6 | 5
  Follow-Up Week 100 | -6.3 (7.20) | -3.9 (4.62)

14. Secondary Outcome: Change From Baseline in the Pericardial/Pleuritic Pain Scale During ATEP by Time Poimt
Description: The pericardial/pleuritic pain scale was scored using numerical values of 1 through 10 with 1 representing 'no pain' and 10 representing 'worst possible pain'. These were self-administered by the participants and gauged the severity of their SLE pain related to pericardial and pleuritic discomfort. Any indication from participants or study assessments, aside from pain, which indicated clinically significant pericardial or pleuritic manifestations of SLE was thoroughly investigated; if clinically significant SLE related complications were found, the participants was to be discontinued from the study and entered into the Observational Follow-up Period and treated appropriately.
Time Frame: Baseline to Weeks 1, 4, 12, 24, 36, 48, 60, 72, 84, 96 and follow-up at Week 100 during the ATEP.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ATEP: Iberdomide 0.3 mg QD | ATEP: Iberdomide 0.6 mg/0.3 mg ALT Days
Number analyzed (Participants) | 9 | 8
Units on a Scale
  Week 1 | -1.0 (2.65) | 0.8 (1.49)
  Week 4: number analyzed (Participants) | 9 | 7
  Week 4 | -0.8 (2.74) | 0.9 (2.01)
  Week 12: number analyzed (Participants) | 9 | 7
  Week 12 | -1.1 (2.67) | 1.3 (2.21)
  Week 24: number analyzed (Participants) | 8 | 5
  Week 24 | -1.0 (2.88) | 0.6 (1.34)
  Week 36: number analyzed (Participants) | 7 | 5
  Week 36 | -0.7 (3.30) | 0.7 (1.57)
  Week 48: number analyzed (Participants) | 7 | 5
  Week 48 | -1.4 (2.99) | 0.9 (2.01)
  Week 60: number analyzed (Participants) | 7 | 5
  Week 60 | -1.1 (3.18) | 1.1 (2.41)
  Week 72: number analyzed (Participants) | 6 | 3
  Week 72 | 0.2 (1.57) | 0.0 (0.00)
  Week 84: number analyzed (Participants) | 6 | 2
  Week 84 | 0.2 (0.98) | 0.0 (0.00)
  Week 96: number analyzed (Participants) | 6 | 1
  Week 96 | -0.2 (0.98) | 0.0 (NA) — NA = Could not be calculated due to the low number of participants with available data.
  Follow-Up Week 100: number analyzed (Participants) | 7 | 5
  Follow-Up Week 100 | -0.6 (0.98) | 0.2 (1.10)

15. Secondary Outcome: Change From Baseline in the Fatigue Visual Analog Scale (VAS) During the ATEP by Time Point
Description: The Fatigue VAS evaluates SLE-related fatigue using a 0 to 100 mm VAS scale. The Fatigue VAS allowed the participant to indicate the degree of SLE-related fatigue by placing an "X" representing how they feel, along a visual analog line that extends between two extremes (e.g., from not at all tired to extremely tired) over the previous week. A decrease in the fatigue VAS indicates improvement.
Time Frame: Baseline to Weeks 1, 4, 12, 24, 36, 48, 60, 72, 84, 96 and follow-up at Week 100 during the ATEP.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ATEP: Iberdomide 0.3 mg QD | ATEP: Iberdomide 0.6 mg/0.3 mg ALT Days
Number analyzed (Participants) | 9 | 8
Units on a Scale
  Week 1 | -10.0 (20.30) | -4.0 (13.48)
  Week 4: number analyzed (Participants) | 9 | 7
  Week 4 | -4.1 (16.96) | -3.7 (12.23)
  Week 12: number analyzed (Participants) | 9 | 7
  Week 12 | -15.9 (30.77) | -8.0 (20.60)
  Week 24: number analyzed (Participants) | 8 | 5
  Week 24 | -13.6 (17.27) | -4.0 (8.80)
  Week 36: number analyzed (Participants) | 7 | 5
  Week 36 | -21.1 (20.96) | -17.2 (17.48)
  Week 48: number analyzed (Participants) | 7 | 5
  Week 48 | -29.9 (20.58) | -12.8 (14.48)
  Week 60: number analyzed (Participants) | 7 | 5
  Week 60 | -23.0 (20.65) | -12.6 (10.74)
  Week 72: number analyzed (Participants) | 6 | 3
  Week 72 | -22.8 (26.96) | -25.7 (19.55)
  Week 84: number analyzed (Participants) | 6 | 2
  Week 84 | -10.3 (24.61) | -14.0 (19.80)
  Week 96: number analyzed (Participants) | 6 | 1
  Week 96 | -9.8 (34.52) | -20.0 (NA) — NA = Could not be calculated due to the low number of participants with available data.

16. Secondary Outcome: Change From Baseline in the Cutaneous Lupus Area and Severity Index (CLASI) Damage Score During the ATEP by Time Point
Description: as for outcome 11
Time Frame: Baseline to Weeks 1, 4, 12, 24, 36, 48, 60, 72, 84, 96 and follow-up at Week 100 during the ATEP.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ATEP: Iberdomide 0.3 mg QD | ATEP: Iberdomide 0.6 mg/0.3 mg ALT Days
Number analyzed (Participants) | 9 | 8
Units on a Scale
  Week 1 | -0.1 (0.33) | 0.0 (0.00)
  Week 4: number analyzed (Participants) | 9 | 7
  Week 4 | 0.0 (0.00) | -1.0 (2.24)
  Week 12: number analyzed (Participants) | 8 | 7
  Week 12 | -0.6 (1.77) | -0.9 (2.73)
  Week 24: number analyzed (Participants) | 8 | 5
  Week 24 | 0.1 (0.83) | -2.2 (4.38)
  Week 36: number analyzed (Participants) | 7 | 5
  Week 36 | 0.1 (0.38) | -2.2 (4.38)
  Week 48: number analyzed (Participants) | 7 | 5
  Week 48 | 0.3 (0.76) | -2.4 (4.83)
  Week 60: number analyzed (Participants) | 7 | 5
  Week 60 | 0.4 (0.79) | -2.6 (5.81)
  Week 72: number analyzed (Participants) | 6 | 3
  Week 72 | 0.3 (0.82) | -0.7 (1.15)
  Week 84: number analyzed (Participants) | 6 | 2
  Week 84 | 0.7 (1.63) | -1.0 (1.41)
  Week 96: number analyzed (Participants) | 6 | 1
  Week 96 | 0.0 (0.00) | 0.0 (NA) — NA = Could not be calculated due to the low number of participants with available data.
  Follow-Up Week 100: number analyzed (Participants) | 7 | 5
  Follow-Up Week 100 | -0.3 (1.25) | 0.0 (0.00)

17. Secondary Outcome: Change From Baseline in the Systemic Lupus International Collaborating Clinics/American College of Rheumatology Systemic Lupus Erythematosus (SLICC/ACR SLE) Damage Index Score During the ATEP by Time Point
Description: SLICC/ACR score or damage index is a measure of cumulative damage due to Systemic Lupus Erythematosus (SLE). Damage is defined as nonreversible change (not related to active inflammation) occurring since onset of lupus, ascertained by clinical assessment and present for at least 6 months. Damage is defined for 12 separate organ systems: ocular (range 0-2), neuropsychiatric (0-6), renal (0-3), pulmonary (0-5), cardiovascular (0-6), peripheral vascular (0-5), gastrointestinal (0-6), musculoskeletal (0-7), skin (0-3), endocrine (diabetes) (0-1), gonadal (0-1) and malignancies (0-2). A score of 0=no damage, early damage is defined as ≥1. The total maximum score is 47, and increasing score indicates increasing disease damage severity.
Time Frame: Baseline to Weeks 1, 4, 12, 24, 36, 48, 60, 72, 84, 96 and follow-up at Week 100 during the ATEP.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | ATEP: Iberdomide 0.3 mg QD | ATEP: Iberdomide 0.6 mg/0.3 mg ALT Days
Number analyzed (Participants) | 9 | 8
Units on a Scale
  Week 1 | -0.1 (0.33) | 0.0 (0.00)
  Week 4: number analyzed (Participants) | 9 | 7
  Week 4 | -0.1 (0.33) | -0.1 (0.38)
  Week 12: number analyzed (Participants) | 8 | 7
  Week 12 | -0.1 (0.35) | -0.1 (0.38)
  Week 24: number analyzed (Participants) | 8 | 5
  Week 24 | -0.1 (0.35) | -0.2 (0.45)
  Week 36: number analyzed (Participants) | 7 | 5
  Week 36 | 0.0 (0.00) | -0.2 (0.45)
  Week 48: number analyzed (Participants) | 7 | 5
  Week 48 | 0.0 (0.00) | -0.2 (0.45)
  Week 60: number analyzed (Participants) | 7 | 5
  Week 60 | 0.0 (0.00) | -0.2 (0.45)
  Week 72: number analyzed (Participants) | 6 | 3
  Week 72 | 0.0 (0.00) | 0.0 (0.00)
  Week 84: number analyzed (Participants) | 6 | 2
  Week 84 | 0.0 (0.00) | 0.0 (0.00)
  Week 96: number analyzed (Participants) | 6 | 1
  Week 96 | 0.0 (0.00) | 0.0 (NA) — NA = Could not be calculated due to the low number of participants with available data.
  Follow-Up Week 100: number analyzed (Participants) | 7 | 5
  Follow-Up Week 100 | 0.6 (1.13) | 0.0 (0.00)

ADVERSE EVENTS:
Time Frame: TEAEs were monitored from the date of the first dose of IP until 28 days after the last dose of IP or study IP discontinuation in Part 1; median treatment duration was 12.0 weeks for the placebo, 0.3 mg Iberdomide QOD and 0.3 mg QD cohorts and 11.9 weeks for the 0.6/0.3 ALT and 0.6 cohorts
Description: For the ATEP, TEAEs were monitored from the date of the first dose of IP until 28 days after the last dose or study IP discontinuation; median duration of treatment was 95.86 weeks for the 0.3 mg iberdomide QD cohort and 60.64 weeks for the 0.6 mg/0.3 mg ALT QD cohorts.
Groups:
- Part 1: Iberdomide 0.6 mg/ 0.3 mg ALT QD: Participants received iberdomide 0.6 mg and 0.3 mg on alternating days for up to 84 days during the Part 1 treatment phase.
- ATEP: Iberdomide 0.6 mg/ 0.3 mg ALT QD: Participants originally randomized to iberdomide 0.6 mg capsules QD or 0.6 mg Iberdomide capsules alternating days with 0.3 mg iberdomide capsules or placebo capsules QD chorts (in these respective groups), during the Part 1 treatment phase, were assigned 0.3 mg iberdomide capsules ALT days with 0.6 mg capsules ALT days when entered into the active treatment extension phase up to 2 years.
Arm/Group | Part 1: Placebo | Part 1: Iberdomide 0.3 mg QOD | Part 1: Iberdomide 0.3 mg QD | Part 1: Iberdomide 0.6 mg/ 0.3 mg ALT QD | Part 1: Iberdomide 0.6 mg QD | ATEP: Iberdomide 0.3 mg QD | ATEP: Iberdomide 0.6 mg/ 0.3 mg ALT QD
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/9 | 0/9 | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 2/8 | 0/8 | 0/8 | 1/9 | 1/9 | 0/9 | 4/8
Other Adverse Events (participants affected / at risk) | 5/8 | 7/8 | 7/8 | 8/9 | 8/9 | 9/9 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo (N=8) | Part 1: Iberdomide 0.3 mg QOD (N=8) | Part 1: Iberdomide 0.3 mg QD (N=8) | Part 1: Iberdomide 0.6 mg/ 0.3 mg ALT QD (N=9) | Part 1: Iberdomide 0.6 mg QD (N=9) | ATEP: Iberdomide 0.3 mg QD (N=9) | ATEP: Iberdomide 0.6 mg/ 0.3 mg ALT QD (N=8)
Vitreous detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Schizoaffective disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo (N=8) | Part 1: Iberdomide 0.3 mg QOD (N=8) | Part 1: Iberdomide 0.3 mg QD (N=8) | Part 1: Iberdomide 0.6 mg/ 0.3 mg ALT QD (N=9) | Part 1: Iberdomide 0.6 mg QD (N=9) | ATEP: Iberdomide 0.3 mg QD (N=9) | ATEP: Iberdomide 0.6 mg/ 0.3 mg ALT QD (N=8)
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Episcleritis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Keratitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ocular discomfort (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Retinopathy hypertensive (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Scleritis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dental necrosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 1 | 2 | 2 | 1 | 3
Duodenal polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lip blister (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 3 | 3 | 0 | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bacteriuria (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 3 | 3
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Herpes virus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lyme disease (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 2 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 1 | 1 | 4 | 3
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 2 | 2
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypovitaminosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nerve root compression (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Small fibre neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Generalised anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Irritability (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Middle insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cervical polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Galactorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nipple disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash follicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is > 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 additional days. Investigator must delete confidential information before submission and defer publication to permit patent applications.

DOCUMENTS (3):
  • Study Protocol (2018-06-18): https://cdn.clinicaltrials.gov/large-docs/40/NCT02185040/Prot_000.pdf
  • Statistical Analysis Plan: CC-220-SLE-001-SAP-Part1_Redacted25July2016 (2016-07-25): https://cdn.clinicaltrials.gov/large-docs/40/NCT02185040/SAP_001.pdf
  • Statistical Analysis Plan: CC-220-SLE-001-ATEP.31Oct2018_Redacted (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/40/NCT02185040/SAP_002.pdf